CLINICAL TRIAL: NCT03826446
Title: Laparoscopic Versus Open Complete Mesocolic Excision With Central Vascular Ligation in Right Colon Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Karim Mohamed Shady, kshady- Principal investigstor, Menoufia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Faculty of medicine-MenoufiaU
Record Dates: First submitted 2019-01-27; First posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Colon Cancer
Keywords: Right colon cancer; Mesocolic excision
MeSH Terms: conditions — Colonic Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Surgery (Other): Patients diagnosed as operable right sided colon cancer were enrolled in this study and did open complete mesocolic excision procedures
  Interventions: Procedure: Surgery
- Laparoscopic Surgery (Other): Patients diagnosed as operable right sided colon cancer were enrolled in this study and did laparoscopic complete mesocolic excision procedures
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — laparoscopic and open complete mesocolic excision with central vascular ligation in right colon cancer.

SUMMARY:
Right sided hemicolectomy is the standard type of operation for cancers in the caecum, the ascending colon.The aim of this study was to compare between laparoscopic and open complete mesocolic excision with central vascular ligation in right colon cancer.

DETAILED DESCRIPTION:
Colorectal cancer incidence and mortality rates vary markedly around the world. Globally, colorectal cancer is the third most commonly diagnosed cancer in males and the second in females, with 1.65 million new cases and almost 835,000 deaths in 2015. Rates are substantially higher in males than in females.

The right colon has a large caliber, a thin wall, and its contents are liquid; thus, obstruction is a late event. Bleeding is usually occult. Fatigue and weakness caused by severe anemia may be the only complaints. Tumors sometimes grow large enough to be palpable through the abdominal wall before other symptoms appear.

Curative treatment for right colon cancer includes resection of the tumor-bearing bowel segment. There are standard types of operations, depending on the location of the tumor. The types of standard resections are based on the knowledge of lymphatic drainage and lymph node anatomy.

Right sided hemicolectomy is the standard type of operation for cancers in the caecum, the ascending colon. In 2009, Hohenberger, a German scholar, proposed the term of complete mesocolic excision (CME), whose basic theory is mainly composed of two concepts in fetal anatomy and surgical oncology: sharp dissection of the mesocolic plane and the parietal plane. CME helps to keep the colonic mesentery intact, clarify the dissected area from central lymph nodes, emphasize the importance of transecting colon-feeding blood at the root, and increase the range of longitudinal enterotomy. Thus, CME provides a standardization of surgeries for colon cancer.

Traditionally, approach to right colon cancer is through open exploration but this approach has more blood loss, prolonged postoperative hospital stay, sever postoperative pain and delayed recovery..

Laparoscopic right colectomy (LRC) for colon cancer became a well-established technique in the surgical armamentarium of colorectal operations. It has well proved advantages: reduction in postoperative pain, time to return of bowel function, and length of hospital stay.

The purpose of the present study was to compare between laparoscopic and open complete mesocolic excision with central vascular ligation in right colon cancer as regards technical feasibility, advantages and disadvantages of both procedures.

This was prospective randomized study and was carried out on 60 patients diagnosed as operable right sided colon cancer and the patients will be divided into two groups:

Group I: Open right hemicolectomy with complete mesocolic excision with central vascular ligation.

Group II: Laparoscopic right hemicolectomy with complete mesocolic excision with central vascular ligation.

All patients were subjected to preoperative assessment in the form of:

* Full history.
* Clinical evaluation and body weight.
* Laboratory investigation (Complete blood picture, liver function tests, blood sugar, blood urea, serum creatinine, prothrombin time, serum albumin and tumour markers(.
* Imaging (chest X-ray, US abdomen, CT abdomen and pelvis).
* Histopathology diagnosis (endoscopic biopsy, tissue diagnosis).

Operative technique

In patients of group I:

* A standard mechanical bowel preparation will be performed 24 hours before operation.
* The patient will be placed in the supine position and the operation will be carried out in a standard manner.
* A midline incision of about 15 to 20 cm will be made.
* The right-sided colon will be mobilized before mesenteric division and the same vessels will be dissected frequently.
* Ileotransverse end-to-end hand anastomosis is operated and the mesenteric defect will be closed.

In patients of group II:

* A standard mechanical bowel preparation will be performed 24 hours before the operation.
* A high-definition laparoscope will be used.
* Under general anaesthesia the operation is carried out in standard manner, with the patient in a modified lithotomy position.
* After achieving pneumoperitoneum (12 mm Hg), a 12-mm trocar will be placed through an incision just above the umbilicus, and a 30-degree laparoscope will be inserted through the 12-mm trocar. The second 10-mm trocar will be inserted at the upper left quadrant of the abdomen for the major acting port. The third 5-mm trocar will be inserted at the lower left quadrant for the second major active port. The fourth and fifth 5-mm trocars will be inserted at the upper right and lower right quadrants.
* According to laparoscopic procedure, the position, composition, and spatial relationships of the surgery planes needed for laparoscopic complete mesocolic excision for right sided colic cancer cases are identified.

Intraoperatively, all patients will be assessed for:

* Time of the procedure.
* Amount of blood loss.

Postoperative follow up:

Patients will be followed up by the standardized follow up protocol. They will be examined by the outpatient setting after:

* 2 weeks (post-operative) for: wound infection, leakage, pathological outcome (The tumor node metastasis (TNM) stage, histologic grade of differentiation, number of harvested lymph nodes, lymphovascular invasion, estimation of resection margins).
* Every 3 months for 1-2 years by: history taking, physical examination, carcinoembryonic antigen measurement,
* Every 6 months for 1-2 years by: chest, abdomen-pelvic computed tomography for detection of local or systemic recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Only operable cases of right colon cancer by (CT scan criteria) which include:

  1. No permeation of surrounding fat planes.
  2. No encasement of major vascular structures.
  3. No extensive local spread.
  4. No distant metastases or peritoneal infiltration were included in this study.

Exclusion Criteria:

* 1- All cases with perforation or obstruction. 2- Metastatic colon cancer. 3- Patients undergoing colectomy including another part of the colon than right colon.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Operative time in open and laparoscopic complete mesocolic excision groups in right cancer colon | 1-3 years
  Comparing the operative time between laparoscopic and open complete mesocolic excision with central artery ligation groups
Incision length in open and laparoscopic complete mesocolic excision groups in right cancer colon | 1-3 years
  Comparing the incision length between laparoscopic and open complete mesocolic excision with central artery ligation groups
Hospital stay duration in open and laparoscopic complete mesocolic excision groups in right cancer colon | 1-3
  Comparing the hospital stay duration between laparoscopic and open complete mesocolic excision with central artery ligation groups
Histopathological findings in open and laparoscopic complete mesocolic excision groups in right cancer colon | 1-3 years
  Comparing the histopathological findings between laparoscopic and open complete mesocolic excision with central artery ligation groups
Post-operative complications in open and laparoscopic complete mesocolic excision groups in right cancer colon | 1-3 years
  Comparing the post-operative complications between laparoscopic and open complete mesocolic excision with central artery ligation groups
Recurrence rate in open and laparoscopic complete mesocolic excision groups in right cancer colon | 1-3 years
  Comparing the recurrence rate between laparoscopic and open complete mesocolic excision with central artery ligation groups

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, ShebinElkom, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided